CLINICAL TRIAL: NCT06767085
Title: Pain Management With Lidocaine-prilocaine Spray During Diagnostic Office Hysteroscopy in Postmenopausal Women: a Randomized Controlled Study
Brief Title: Pain Management During Diagnostic Office Hysteroscopy in Postmenopausal Women: a Randomized Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP SPRAY HYSTEROSCOPY
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Office Hysteroscopy
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine prilocaine (Experimental)
  Interventions: Drug: Lidocaine-Prilocaine Topical
- placebo (Placebo Comparator)
  Interventions: Drug: Saline spray

INTERVENTIONS:
Drug: Lidocaine-Prilocaine Topical — lidocaine-prilocaine spray on the cervix and cervical canal 5-7 minutes prior to the procedure
  Arms: lidocaine prilocaine
Drug: Saline spray — saline spray on the cervix and cervical canal 5-7 minutes prior to the procedure
  Arms: placebo

SUMMARY:
To assess the effectiveness of lidocaine-prilocaine spray versus placebo in minimizing the pain experienced by postmenopausal patients during diagnostic ofﬁce hysteroscopy and to assess the ease of insertion of hysteroscope as reported by the hysteroscopists

DETAILED DESCRIPTION:
To assess the effectiveness of lidocaine-prilocaine spray versus placebo in minimizing the pain experienced by postmenopausal patients during diagnostic ofﬁce hysteroscopy and to assess the ease of insertion of hysteroscope as reported by the hysteroscopists

ELIGIBILITY:
Inclusion Criteria:

* Menopausal patients with an indication for ofﬁce hysteroscopy (postmenopausal bleeding or abnormal ultrasound ﬁndings)

Exclusion Criteria:

* Nulliparous patients patients with cervical pathology retroverted uterus (detected by transvaginal ultrasound) previous cervical surgery patients with severe vaginal bleeding allergy or contraindications to lidocaine-prilocaine spray

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-02-05 (Estimated); Primary Completion 2025-07-05 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain | 5 minutes
  Pain intensity will be assessed by visual analogue scale during the procedure.visual analogue scale ranging from 0 to 10

SECONDARY OUTCOMES:
Intensity of pain | 20 minutes
  Pain intensity will be assessed by visual analogue scale 30 minutes after the procedure.visual analogue scale ranging from 0 to 10
ease of insertion | 5 MINUTES
  ease of insertion by 10 CM VAS LIKE SCORE in which 10 means terribly difficult entry and 0 means very easy entry

IPD SHARING:
Plan to Share IPD: Undecided